CLINICAL TRIAL: NCT01831128
Title: Prospective Multicentre Observational French Cohort Study of Patients With Heart Failure and Central Sleep Apnoea Requiring Adaptive Servo-Ventilation (PaceWave, AutoSet CS) Treatment
Brief Title: French Cohort Study of Chronic Heart Failure Patients With Central Sleep Apnoea Eligible for Adaptive Servo-Ventilation (PaceWave, AutoSet CS)
Acronym: FACE
Status: Completed | Type: Observational
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: FACE 001
Record Dates: First submitted 2013-04-02; First posted 2013-04-15 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Chronic Heart Failure; Central Sleep Apnea
Keywords: Congestive Heart Failure; Central Sleep Apnea; Sleep-Disordered Breathing
MeSH Terms: conditions — Sleep Apnea, Central; Heart Failure; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ASV Treatment: AutoSet CS, PaceWave
  Interventions: Device: ASV Treatment
- Control: No ASV treatment

INTERVENTIONS:
Device: ASV Treatment
  Other Names: PaceWave; AutoSet CS
  Groups: ASV Treatment

SUMMARY:
The purpose of FACE study is to provide in routine practice complementary long-term data on the mortality and morbidity of Chronic Heart Failure (CHF) patients with Central Sleep Apnea eligible for Adaptative Servo-Ventilation (ASV) treatment (PaceWave, AutoSet CS; ResMed).

DETAILED DESCRIPTION:
The prevalence of Central Sleep Apnea (CSA) and/or Cheyne-Stokes Respiration (CSR) in patients with Chronic Heart Failure (HF) is 15-46% and it is associated with worse prognosis. Adaptative Servo-Ventilation (ASV) suppresses sleep apnoea and reduces hyperventilation, and is more effective than continuous positive airway pressure (CPAP) for treating CSA/CSR. Short-term studies show that ASV improves cardiac function and quality of life in CHF patients.

The SERVE HF multinational randomized trial is assessing the effects of addition of ASV (PaceWave, AutoSet CS; ResMed) to optimal medical management compared with medical management alone in symptomatic CHF patients with altered Left Ventricular Ejection Fraction and predominant CSA/CSR. The FACE study is a French prospective, multicentre, observational cohort that will provide complementary data to SERVE HF trial by characterizing CHF population eligible for ASV indications and evaluating the treatment management on long term follow-up of CHF patients with CSA/CSR in routine practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patient with Chronic Heart Failure
* Central Sleep Apnea requiring ASV therapy

Exclusion Criteria:

* Contra-indications to ASV therapy
* Respiratory Failure or Hypercapnia inconsistent with ASV therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Heart Failure Patients with Central Sleep Apnea
Sampling Method: Non-Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Time to first event of all cause mortality or unplanned hospitalization for worsening heart failure | 2 years
Time to first event of cardiovascular mortality or unplanned hospitalization for worsening heart failure | 2 years
Time to first event of all cause mortality or all cause hospitalization | 2 years

SECONDARY OUTCOMES:
Time until death | 2 years
Time to non cardiovascular death | 2 years
Time to cardiovascular death | 2 years
Time to hospitalization due to deterioration of heart failure or cardiovascular death | 2 years
Time to hospitalization for other reasons or death | 2 years
Time to hospitalization for cardiovascular cause or cardiovascular death | 2 years
Changes in CHF stage by evaluating NYHA (New York Heart Association) class as compared to baseline | 2 years
Changes in Quality Of Life by measuring Minnesota score as compared to baseline | 2 years
Changes in LVEF (Left Ventricular Ejection Fraction) as compared to baseline | 2 years
Changes in Heart Rhythm as compared to baseline | 2 years
Changes in Systolic and diastolic Blood Pressure | 2 years
Changes in AHI (Apnea Hypopnea Index) as compared to baseline | 2 years
Changes in renal function as compared to baseline | 2 years
  Estimated GFR (eGFR) will be calculated using the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) formula
Changes in BNP (B-type Natriuretic Peptide) rates as compared to baseline | 2 years
Changes in Daytime Sleepiness by measuring Epworth scale as compared to baseline | 2 years
ASV Compliance | 2 years
Changes in medical treatment as compared to baseline | 2 years
  Medication consumption and use of cardiac implant will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pia d'ORTHO, MD, PhD, Principal Investigator — APHP (Assistance Publique Hôpitaux de Paris) - Bichat-Claude Bernard Hospital, Paris; Jean-Louis PEPIN, MD, PhD, Study Chair — Grenoble University Hospital, Grenoble; Jean-Marc DAVY, MD, PhD, Study Chair — Arnaud de Villeneuve University Hospital, Montpellier; Thibaud DAMY, MD, PhD, Study Chair — APHP - Henri Mondor University Hospital, Creteil; Patrick LEVY, MD, PhD, Study Chair — Grenoble University Hospital, Grenoble; Renaud TAMISIER, MD, PhD, Study Chair — Grenoble University Hospital, Grenoble
Locations (18):
- France (18):
  - Medical practice of cardiology, Amnéville
  - Angers University Hospital, Angers
  - Antibes Hospital, Antibes
  - Béziers Hospital, Béziers
  - Cannes Hospital, Cannes
  - Henri-Mondor University Hospital, Créteil
  - Grenoble University Hospital, Grenoble
  - Le Mans Hospital, Le Mans
  - HCL - Croix-Rousse Hospital, Lyon
  - Jacques Cartier Hospital, Massy
  - Arnaud de Villeneuve University Hospital, Montpellier
  - Nevers Hospital, Nevers
  - APHP - Pitié-Salpêtrière University Hospital, Paris
  - APHP - Bichat-Claude Bernard Hospital, Paris
  - Bordeaux University Hospital, Pessac
  - Poitiers University Hospital, Poitiers
  - Saint Laurent Polyclinic, Rennes
  - Toulouse University Hospital, Toulouse

REFERENCES:
- [Derived] Tamisier R, Damy T, Bailly S, Goutorbe F, Davy JM, Lavergne F, Palot A, Verbraecken JA, d'Ortho MP, Pepin JL; FACE investigators; Steering committee members; d'Ortho MP, Pepin JL, Davy JM, Damy T, Tamisier R; FACE study investigators. FACE study: 2-year follow-up of adaptive servo-ventilation for sleep-disordered breathing in a chronic heart failure cohort. Sleep Med. 2024 Jan;113:412-421. doi: 10.1016/j.sleep.2023.07.014. Epub 2023 Jul 22. PMID 37612192
- [Derived] Tamisier R, Damy T, Davy JM, Verbraecken JA, Bailly S, Lavergne F, Palot A, Goutorbe F, Pepin JL, d'Ortho MP. Cohort profile: FACE, prospective follow-up of chronic heart failure patients with sleep-disordered breathing indicated for adaptive servo ventilation. BMJ Open. 2020 Jul 19;10(7):e038403. doi: 10.1136/bmjopen-2020-038403. PMID 32690535